CLINICAL TRIAL: NCT01014156
Title: Effects of Intravenous Epoprostenol Sodium (Flolan®) in Patients With Moderate-to-Severe Pulmonary Thrombo-Embolism
Brief Title: Epoprostenol in Pulmonary Embolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Free University Medical Center (Other)
Responsible Party: Albertus Jozef Kooter, Free University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03.123
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Acute Pulmonary Embolism
Keywords: pulmonary embolism; vasoconstriction; right ventricular dysfunction; epoprostenol; acute pulmonary embolism with right ventricular dysfunction
MeSH Terms: conditions — Pulmonary Embolism; Ventricular Dysfunction, Right | interventions — Epoprostenol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- epoprostenol intraveneously (Experimental): epoprostenol iv versus placebo iv, both on top of low molecular weight heparin
  Interventions: Drug: epoprostenol

INTERVENTIONS:
Drug: epoprostenol — titration up to 4 ng/kg/min
  Other Names: prostacyclin, flolan

SUMMARY:
You are admitted to hospital because of pulmonary embolism. You are treated with anticoagulants.

The investigators know that, despite this treatment, pulmonary embolism can be a threat especially if heart function is compromized.

The investigators investigate a well known study drug (epoprostenol) on top of regular treatment with anticoagulants, to see if heart function can be optimized

DETAILED DESCRIPTION:
Pulmonary thromboembolism (PE) with circulatory and/or respiratory symptoms is associated with high morbidity and mortality. Acute pulmonary hypertension is the hallmark of severe PE, and is to be held responsible for the full spectrum of clinical manifestations and complications. Although it is common belief that only mechanical obstruction by thrombus mass causes this pulmonary hypertension, there is strong evidence indicating that pulmonary vasoconstriction contributes significantly to the rise in pulmonary vascular resistance.

Although all patients will receive anticoagulant treatment immediately after the diagnosis is established, morbidity and mortality are still disturbingly high when circulatory and/or respiratory symptoms accompany PE, or when hemodynamically stable PE patients have echocardiographic signs of acute right ventricle overload. There are no generally accepted guidelines for additional treatment options in these patients with moderate-to-severe PE. Thrombolytic therapy is recommended by many when hemodynamic symptoms are severe, but its effectiveness has never been proven in a controlled trial. In patients with moderate-to-large PE associated with echocardiographic signs of right ventricle overload, but who are still circulatory stable, mortality is increased, but thrombolytic therapy appears not to be beneficial.

Given the plausible role of pulmonary vasoconstriction in the pathogenesis of PE associated pulmonary hypertension, the potential benefit of pulmonary vasodilators is important.There is experimental evidence that antagonising pulmonary vasoconstriction by the administration of selective vasodilators may be beneficial in animals with PE. In addition, anecdotal evidence of a similar kind exists for humans with acute PE.

We hypothesise that in PE patients who have echocardiographic evidence of acute right ventricle overload, epoprostenol sodium (Flolan®) results in partial or complete reversal of echocardiographic abnormalities, as well as in improvement in respiratory and circulatory symptoms and signs.

ELIGIBILITY:
Inclusion Criteria:

* acute (symptoms <24 hrs) with right ventricular dilatation (>30 mm end diastolic, systolic PAP > 50 mmHg,
* absence of right ventricular wall hypertrophy)

Exclusion Criteria:

* age below 18 years or above 70 years
* body mass index >35 kg/m2
* duration of symptoms >24 hours (since onset or acute increase in symptoms)
* severe circulatory shock (systemic blood pressure systolic <80 mmHg, or diastolic blood pressure <45 mmHg) or respiratory failure, requiring mechanical ventilation.
* patients who, in the opinion of the supervising physician, require thrombolytic therapy.
* severe pre-existent cardiopulmonary disease (heart failure, obstructive pulmonary disease, emphysema)
* atrial fibrillation
* refusal or inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Right ventricular end diastolic diameter (ultrasound) | 0, 2,5 4, 24 and 72 hours

SECONDARY OUTCOMES:
systolic pulmonary artery pressure (ultrasound) | identical to primary measure

CONTACTS AND LOCATIONS:
Locations (1):
- Free University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Kooter AJ, Ijzerman RG, Kamp O, Boonstra AB, Smulders YM. No effect of epoprostenol on right ventricular diameter in patients with acute pulmonary embolism: a randomized controlled trial. BMC Pulm Med. 2010 Mar 30;10:18. doi: 10.1186/1471-2466-10-18. PMID 20353588